CLINICAL TRIAL: NCT00427271
Title: Aspirin and the Antiproteinuric Effect of Enalapril in Microalbuminuric Type 2 Diabetes Mellitus Patients: a Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Aspirin and Enalapril in Microalbuminuric Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02-353
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes Mellitus; Microalbuminuria
Keywords: aspirin; enalapril; microalbuminuria; glomerular filtration rate
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aspirin

INTERVENTIONS:
Drug: aspirin

SUMMARY:
Research design: randomized, double-blind, placebo-controlled crossover study to evaluate the putative interference of low-dose aspirin (for 8 weeks) on enalapril antiproteinuric properties in microalbuminuric type 2 diabetes mellitus patients

DETAILED DESCRIPTION:
Research design: randomized, double-blind, placebo-controlled crossover study Patients: Microalbuminuric (urinary albumin excretion [UAE]30-300 mg/d)type 2 diabetes mellitus patients without ischemic heart disease or peptic ulcer Aim:To evaluate the putative interference of low-dose aspirin (300 mg/d)for 8 weeks)on enalapril antiproteinuric properties in microalbuminuric type 2 diabetes mellitus patients Study protocol:Crossover randomization to 8 weeks of enalapril 10 mg/d plus aspirin (300 mg/d) or plus placebo, and a 6-week washout period. Measurement of UAE (immunoturbidimetry) and glomerular filtration rate (51Cr-EDTA), blood pressure and metabolic control at baseline and at the end of each period.

Statistical analyses: Bland&Altman analyses for crossover trials.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus microalbuminuria

Exclusion Criteria:

* ischemic heart disease peptic disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-03; Study Completion 2007-01

PRIMARY OUTCOMES:
urinary albumin excretion
glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo G Camargo, Study Director — Programa de Pós-graduação em Ciências Médicas: Endocrinologia
Locations (1):
- Hospital de Clínicas de Porto Aelgre, Porto Alegre, Rio Grande do Sul, Brazil